CLINICAL TRIAL: NCT05903261
Title: Prospective Observational Basket Study of Stereotactic Body Radiation Therapy for OligoMetastatic Patients From Rare Tumors: the PROMPT Study
Brief Title: Prospective Observational Basket Study of Stereotactic Body Radiation Therapy for OligoMetastatic Patients From Rare Tumors
Acronym: PROMPT
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 3497
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Oligometastatic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Radiation: SBRT — stereotactic body radiation therapy (SBRT)

SUMMARY:
This prospective observational study aims to investigate the effectiveness and safety of SBRT in the management of oligometastases from rare tumors. In addition, the study aims to identify potential differences in treatment efficacy and toxicity between different types of cancer and to provide valuable information on the use of SBRT in these contexts, potentially leading to better treatment options and outcomes for these patients.

DETAILED DESCRIPTION:
Oligometastases, defined as limited number of metastases (commonly from one up to five), are increasingly recognized as a distinct clinical entity in cancer management. Recently, the collaboration of experts from ESTRO and EORTC societies elaborated a consensus document and recommended a classification of oligometastatic patients into specific subcategories, according to 17 disease characterization factors and 5 different questions. Emerging evidence suggests that local treatment of oligometastases with stereotactic body radiation therapy (SBRT) can achieve excellent local control with minimal toxicity.

Indeed, the majority of clinical trials investigating the use of SBRT for oligometastases have focused on common solid tumors. There is limited data on the use of SBRT for oligometastases from rare primary tumors such as melanoma, soft tissue sarcoma, head-neck tumors, gynaecological tumors, Merkel cell carcinoma, thymic carcinoma, gastrointestinal stromal tumors (GIST) and urothelial tumors. Additionally, patients with rare tumors often have limited treatment options, and thus, the use of metastases-directed SBRT may provide a potential curative treatment option for these patients.

The use of SBRT for oligometastases from rare tumors is promising, as local control rates have been reported to be high, and the toxicity profile favorable. Additionally, patients with rare tumors often have limited treatment options, and thus, the use of metastases-directed SBRT may provide a potential curative treatment option for these patients. By investigating multiple rare tumor types within one trial, this study aims to identify potential differences in treatment efficacy and toxicity among the different tumor types, and to provide valuable insights into the use of SBRT in this setting, potentially leading to improved treatment options and outcomes for these patients.

ELIGIBILITY:
Inclusion Criteria:

* ECOG PS 0 - 2
* histologically confirmed diagnosis of rare solid tumors including melanoma, soft tissue sarcoma, head-neck tumors, gynaecological tumors, Merkel cell carcinoma, thymic carcinoma, gastrointestinal stromal tumors (GIST) and urothelial tumors
* No limit to the number of metastases treated with SBRT but all active lesions must be treated with radical intent (primary tumor and metastases)
* Synchronous and metachronous oligometastases, as well as oligorecurrent and oligoprogressive disease are allowed
* Ablative dose intended as a minimum dose of 50Gy EQD2/10 in a maximum of 10 fractions
* No restrictions to prior or on-going systemic therapies

Exclusion Criteria:

* prior treatment with radiation to the same metastatic site
* inability to provide informed consent
* contraindications to SBRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent stereotactic body radiation therapy (SBRT) for oligometastases from rare solid tumors including melanoma, soft tissue sarcoma, head-neck tumors, gynaecological tumors, Merkel cell carcinoma, thymic carcinoma, gastrointestinal stromal tumors (GIST) and urothelial tumors
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
local control of treated metastases at 2 years after SBRT | 2 years
  local control of treated metastases at 2 years after SBRT

SECONDARY OUTCOMES:
overall survival | 2 years
  overall survival
progression-free survival | 2 years
  time for which the patient has no trace oligometastatic progression
distant control | 2 years
  analyze the formation of new metastases distant from the oligometastatic site
toxicity rates | 2 years
  toxicity values caused by SBRT
quality of life of patients | 2 years
  will also be assessed using validated patient-reported outcome measures

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No